CLINICAL TRIAL: NCT07136324
Title: Safety and Efficacy of Endoscopic Ultrasound (EUS) Guided Radiofrequency Ablation (RFA) in the Treatment of Pancreatic Lesions: A Prospective Registry
Brief Title: Safety and Efficacy of EUS-RFA in the Treatment of Pancreatic Lesions: A Prospective Registry
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nirav C Thosani, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-18-0192
Record Dates: First submitted 2021-01-08; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cyst
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Serum and fixed tissues samples (biopsy tissue samples embedded in paraffin).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with pancreatic lesions: Patients with pancreatic lesions undergoing EUS-guided RFA treatment. Patients of either gender that are 18 years of age or older.
  Interventions: Device: EUS-guided RFA treatment

INTERVENTIONS:
Device: EUS-guided RFA treatment — A 19-gauge EUS-RFA catheter will be inserted into pancreatic lesions under EUS guidance. RFA energy is then applied in 2-10 cycles with each cycle lasting about 10-30 seconds and the power setting ranging from 10-30 Watts.

SUMMARY:
Purpose: The purpose of this registry is to track the clinical outcomes and progression of patients with pancreatic lesions receiving endoscopic ultrasound (EUS)-based radiofrequency ablation (RFA) therapy.

Research Design: This study is a 7-year, single-center prospective registry study with annual follow up. Patients with pancreatic lesions undergoing EUS-guided RFA treatment will be studied. There will be no deviation from standard of care procedures.

Procedures to be Used: Following recruitment into the program, eligible patients will undergo EUS-RFA for the treatment of their pancreatic lesion and/or malignancy as part of their standard of care.

Endoscopic Intervention: The EUS-guided intervention will be performed based on a clinical decision. The data will be collected for research purposes. Briefly, the procedure involves advancing a 19-gauge EUS-RFA catheter into the target lesion under EUS-guidance. RFA energy is then applied in 2-10 cycles with each cycle lasting about 10 to 30 seconds and the power setting ranging from 10 to 30 Watts. The same physician who performs the initial EUS-RFA procedure will be responsible for subsequent EUS-RFA procedures.

Risks and Potential Benefits: This is a minimal-risk study with associated physical risks being those part of routine standard of care. Additional risks associated with this study include the possible loss of confidentiality if the patient data or information is inadvertently disclosed outside of this study, risks associated with obtaining blood samples, and risks associated with obtaining tissue samples via biopsy. However, all information will be kept strictly confidential and will be used only for research purposes by the listed investigators. Patients will not receive any additional benefit from the study aside from those received as part of standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of any pancreatic premalignant lesion and/or pancreatic malignancy

Exclusion Criteria:

1. Patients with co-existing malignancies of other organs (or a prior history of such)
2. Patients unable to provide informed consent
3. Patients unable to complete follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are undergoing EUS-RFA for the treatment of their pancreatic lesion(s).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Technical success of the tumor treatment | From the date of patients' index EUS-RFA procedure to the end of their follow-up period at 3 years.
  The efficacy of EUS-RFA in inducing the remission of functional, pre-malignant, and/or malignant solid/cystic pancreatic lesions.

SECONDARY OUTCOMES:
Post-procedure complications observed within 30 days | From the date of patients' EUS-RFA procedure to 30 days following the procedure.
  This will be measured based on the grade of the adverse event (ranging from grade 1 (mild) to grade 5 (death). Some notable adverse events include any deaths, life-threatening complications, congenital anomalies, complications that require intervention to prevent permanent impairment/damage, and hospitalization.
Reduction in the size of the tumor | From the date of patients' index EUS-RFA procedure to the end of their follow-up period at 3 years.
  Cross-sectional imaging will be used to evaluate the size of the pancreatic lesions post-RFA treatment. The tumor length, width, and height in centimeters will be assessed. The dimensions of the largest cyst in centimeters (if there are any cystic components) will also be assessed.
Reduction in systemic tumor markers | From the date of patients' index EUS-RFA procedure to the end of their follow-up period at 3 years.
  Clinically indicated tumor marker assays (CEA, CA 19-9, CA 125, CD40, TNF-α, CD40L) will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Nirav C Thosani, MD, MHA, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Varshney S, Sewkani A, Sharma S, Kapoor S, Naik S, Sharma A, Patel K. Radiofrequency ablation of unresectable pancreatic carcinoma: feasibility, efficacy and safety. JOP. 2006 Jan 11;7(1):74-8. PMID 16407624
- [Background] Ierardi AM, Lucchina N, Bacuzzi A, Marco de C, Bracchi E, Cocozza E, Dionigi G, Tsetis D, Floridi C, Carrafiello G. Percutaneous ablation therapies of inoperable pancreatic cancer: a systematic review. Ann Gastroenterol. 2015 Oct-Dec;28(4):431-9. PMID 26424487
- [Background] Evrard S, Menetrier-Caux C, Biota C, Neaud V, Mathoulin-Pelissier S, Blay JY, Rosenbaum J. Cytokines pattern after surgical radiofrequency ablation of liver colorectal metastases. Gastroenterol Clin Biol. 2007 Feb;31(2):141-5. doi: 10.1016/s0399-8320(07)89344-4. PMID 17347620
- [Background] Haen SP, Pereira PL, Salih HR, Rammensee HG, Gouttefangeas C. More than just tumor destruction: immunomodulation by thermal ablation of cancer. Clin Dev Immunol. 2011;2011:160250. doi: 10.1155/2011/160250. Epub 2011 Dec 29. PMID 22242035
- [Background] Goldberg SN. Radiofrequency tumor ablation: principles and techniques. Eur J Ultrasound. 2001 Jun;13(2):129-47. doi: 10.1016/s0929-8266(01)00126-4. PMID 11369525
- [Background] Yoon WJ, Brugge WR. Endoscopic ultrasonography-guided tumor ablation. Gastrointest Endosc Clin N Am. 2012 Apr;22(2):359-69, xi. doi: 10.1016/j.giec.2012.04.017. PMID 22632957
- [Background] Winter JM, Cameron JL, Campbell KA, Arnold MA, Chang DC, Coleman J, Hodgin MB, Sauter PK, Hruban RH, Riall TS, Schulick RD, Choti MA, Lillemoe KD, Yeo CJ. 1423 pancreaticoduodenectomies for pancreatic cancer: A single-institution experience. J Gastrointest Surg. 2006 Nov;10(9):1199-210; discussion 1210-1. doi: 10.1016/j.gassur.2006.08.018. PMID 17114007
- [Background] Vincent A, Herman J, Schulick R, Hruban RH, Goggins M. Pancreatic cancer. Lancet. 2011 Aug 13;378(9791):607-20. doi: 10.1016/S0140-6736(10)62307-0. Epub 2011 May 26. PMID 21620466